CLINICAL TRIAL: NCT01049958
Title: Prevalence of Patient Ventilator Asynchrony in Trauma and Surgical Patients
Brief Title: Study to Measure the Prevalence of Asynchrony In Mechanically Ventilated Patients
Acronym: Asynchrony
Status: Completed | Type: Observational
Sponsor: University of Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: Robinson-2009-01
Record Dates: First submitted 2010-01-13; First posted 2010-01-15 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2013-01

CONDITIONS: Patient/Ventilator Asynchrony
Keywords: asynchrony; mechanical ventilation; blunt trauma
MeSH Terms: conditions — Patient-Ventilator Asynchrony; Wounds, Nonpenetrating

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will examine the prevalence of patient-ventilator asynchrony and its determinants. Mechanically ventilated trauma patients often experience asynchrony when their pattern of breathing does not match the triggering of a mechanical ventilator.

Asynchrony is thought to be more common in delirious patients, patients with chronic lung disease and those who are heavily sedated. The study will examine the relationship between (1) delirium and sedation and (2) the prevalence of asynchrony in trauma patients.

DETAILED DESCRIPTION:
This is a prospective observational study to determine the prevalence of patient/ventilator asynchrony in a cohort of trauma and surgical patients. There will be two 20-minute periods of observation. The first will be during the first 24 hours of mechanical ventilation and the second will take place when the patient is being weaned from the ventilator and is triggering half or more of all ventilator breaths.

The study team will use computer-captured waveforms to determine the proportion of all breaths that are asynchronous. This proportion is the primary outcome variable of the study.

The study hypothesis is that the proportion of asynchronous breaths is higher in patients with higher levels of sedation, as measured by the Richmond Agitation-Sedation Scale (RASS) and the Confusion Assessment Methods for the Intensive Care Unit (CAM-ICU). This hypothesis will be tested using repeated measures analysis of variance.

ELIGIBILITY:
Inclusion Criteria:

* Trauma or surgical diagnosis
* Patients requiring mechanical ventilation

Exclusion Criteria:

* Patients with no spontaneous breathing efforts due to injury or chemical paralysis
* Patients with leaks in the patient ventilator system precluding evaluation of waveforms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the Surgical and Neurosurgical Intensive Care Units at University Hospital, Cincinnati, OH, who require mechanical ventilation and are aged 18 years or older.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2009-07; Primary Completion 2010-05 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Proportion of asynchronous breaths | 20 minutes during first 24 hours on ventilation and 20 minutes during weaning phase

CONTACTS AND LOCATIONS:
Overall Officials: Bryce Robinson, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University Hospital, Cincinnati, Ohio, United States

REFERENCES:
- [Background] Thille AW, Rodriguez P, Cabello B, Lellouche F, Brochard L. Patient-ventilator asynchrony during assisted mechanical ventilation. Intensive Care Med. 2006 Oct;32(10):1515-22. doi: 10.1007/s00134-006-0301-8. Epub 2006 Aug 1. PMID 16896854
- [Background] Fabry B, Guttmann J, Eberhard L, Bauer T, Haberthur C, Wolff G. An analysis of desynchronization between the spontaneously breathing patient and ventilator during inspiratory pressure support. Chest. 1995 May;107(5):1387-94. doi: 10.1378/chest.107.5.1387. PMID 7750336
- [Background] Nava S, Bruschi C, Fracchia C, Braschi A, Rubini F. Patient-ventilator interaction and inspiratory effort during pressure support ventilation in patients with different pathologies. Eur Respir J. 1997 Jan;10(1):177-83. doi: 10.1183/09031936.97.10010177. PMID 9032512
- [Derived] Robinson BR, Blakeman TC, Toth P, Hanseman DJ, Mueller E, Branson RD. Patient-ventilator asynchrony in a traumatically injured population. Respir Care. 2013 Nov;58(11):1847-55. doi: 10.4187/respcare.02237. Epub 2013 Mar 19. PMID 23513248